CLINICAL TRIAL: NCT02922205
Title: Assessing the Safety and Performance of the Endoscopic Linear Cutter Stapler in Laparoscopic Gastric Bypass Surgery.
Brief Title: Stapler Post-market Observational Study
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-01
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RYGB surgery: Obese patients eligible for laparoscopic Roux-en-Y gastric bypass (RYGB) surgery.
  Interventions: Device: Endoscopic Linear Cutter Stapler and reloads

INTERVENTIONS:
Device: Endoscopic Linear Cutter Stapler and reloads — Endoscopic Linear Cutter Stapler and reloads

SUMMARY:
The purpose of this observational study is to evaluate the safety and performance of the Endoscopic Linear Cutter Stapler and reloads from Fengh Medical used in laparoscopic Roux-en-Y gastric bypass surgery to create anastomoses. The goal of the study will be achieved by assessing the device performance and reporting of peri- and postoperative complications in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

* Age at study entry is at least 18 years.
* Patient must sign and date the informed consent form prior to the index-procedure.
* Patient has a BMI ≥ 35 kg/m with one or more related co-morbidity.
* Patient has a BMI ≥ 40 kg/m.

Exclusion Criteria:

* Patient is pregnant.
* History of bariatric surgery.
* Patient is known to be, or suspected of being unable to comply with the study protocol or proposed follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients eligible for laparoscopic Roux-en-Y gastric bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events related to the index-procedure. | 1 month follow-up
  Determination of postoperative anastomotic leaks and intraluminal/intraperitoneal bleeding.
Number of patients with adverse events related to the index-procedure. | 6 months follow-up
  Determination of postoperative anastomotic leaks and intraluminal/intraperitoneal bleeding.

SECONDARY OUTCOMES:
Number of adverse device effects. | 1, 6, 12 and 24 month follow-up
  Determination of staple line disruption.
Number of patients with bariatric surgery related re-interventions. | 1, 6, 12 and 24 month follow-up
Percentage of excess weight loss. | 1, 6, 12 and month follow-up
  pre-operative weight (kg) minus postoperative weight (kg) divided by the ideal body weight (kg).
Questionnaire on food tolerance. | 1, 6, 12 and 24 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verhelst, Dr., Principal Investigator — ZOL, Genk
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No